CLINICAL TRIAL: NCT03116100
Title: Clinical Situations Leading to the Prescription of Neuroleptics by General Practitioner in the Elderly. Practice Survey
Acronym: NEUGERPRAT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-44 Dr Deschasse
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Behavior Disorders; Neuroleptic
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Behavioral disorders of psychiatric or neurological origin in the elderly are an emerging public health problem. Its management can include a prescription of psychotropic drugs (anxiolytics, hypnotics, neuroleptics, antidepressants for the most part). Many studies highlight the misuse of psychotropic drugs in this specific and vulnerable population, as well as the need for targeted actions.

As for neuroleptics, there is a deleterious over-prescription in the so-called productive behavioral disorders (cries, agitation, aggressiveness, ambulation), in particular in the patient with Alzheimer's disease (80% of patients) or related. The same applies to behavioral disorders in an acute episode of confusion, which also constitute a situation for the prescribing of psychotropic drugs in the elderly. The frailty of the elderly associated with neuroleptics is the cause of a significant iatrogenic (falls, confusions, excessive sedation, etc.), iatrogeny is largely avoidable.

There is little data on the representation of behavioral disorders in the elderly, whereas the recognition and management of behavioral disorders are functions of the tolerance of the entourage and the training of the caregivers. Significant data exist in the literature about diagnosis, risk factors, factors favoring or triggering behavioral disorders and somatic pathologies to be sought urgently.

The available recommendations on the drug treatment of behavioral disorders are complex and inappropriate in light of new data, including the dangerousness of psychotropic drugs. The deleterious effect of long-term drug treatments is proved. There is no validated drug strategy, especially in acute confusions of the elderly.

One study showed that there was a change in the type of neuroleptic prescribed between 2003 and 2010. Half of the general practitioners studied during this period switched from a first-generation neuroleptic to a second-generation neuroleptic. Nevertheless, the type of molecule chosen remains at the discretion of the treating physician or even required a psychiatric opinion or a passage in the emergencies. In the case where the practitioner initiates a prescription in office, in the home or in EHPAD, certain situations require the choice of a neuroleptic with or without pre-therapeutic assessment.

ELIGIBILITY:
Inclusion Criteria:

* General practitioner of the Somme,
* Having patients aged 75 and over

Exclusion Criteria:

* General practitioner with a complementary specialty related to psychiatry, neurology or geriatrics (capacity, university degree or inter-university)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Describe the prescription of neuroleptics in patients aged 75 years or older in 2016 in chronic hallucinatory psychosis, behavioral disorders in dementia and confusional outpatient syndrome in general practitioners in the Somme
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Analyzes of the questionnaires on professional practices in patients aged 75 years | 1 day
  Analyzes of the questionnaires on professional practices in patients aged 75 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France